CLINICAL TRIAL: NCT01458860
Title: Aortic Calcification - is it a Marker for Carotid Artery Stenosis?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ZIV-11-0041
Record Dates: First submitted 2011-10-24; First posted 2011-10-25 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Carotid Artery Stenosis; Aortic Calcification
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GROUP A: patients had a CT
- GROUP B: patients with severe carotid artery stenosis

SUMMARY:
Atherosclerosis is the major contributor for the morbidity and mortality for the variety of cardiovascular diseases.

Aortic calcification on x-ray is a marker for arterial atherosclerosis and an independent prognostic factor for the morbidity and mortality from a cardiovascular event.

Carotid artery stenoses is the current accepted indication for interventional treatment of carotid artery, for the prevention of embolic event, while other arterial atherosclerosis indication, is for hemodynamic disturbance and ischemic outcome.

This research will try to find whether incidental aortic calcification can predict carotid artery stenosis.

Two groups will be chosen: group A - patients who had CT scan in the hospital (for different indications); Group B - patients (not from the first group) who have a significant carotid artery stenosis who are indicated for interventional treatment.

The data to analyze:

Group A - Patients with aortic calcification, carotid artery stenosis, and patients with both Group B - Patients who have aortic calcification Comparison of the populations within the group and among the two will show if a significant correlation between aortic calcification and carotid artery stenosis exist.

DETAILED DESCRIPTION:
Background - thoracic or abdominal aortic calcification is a documented independent risk factor for cardiovascular atherosclerotic disease and increased death.

Atherosclerosis is a diffuse multicentric disease in the arterial tree, affecting target organs (heart, aorta, lower extremities, carotid arteries etc.). Mostly located in arterial bifurcations (Iliac and carotid artery bifurcations) or in constant repetitive arterial trauma (Adductors tendon, Hunter's canal). The invasive treatment (endovascular, surgery) is preserved for patients with critical arterial stenosis or occlusion in symptomatic patients. Exceptions are the carotid arteries: the majority of patients with a severe internal carotid artery stenosis are asymptomatic patients, which are treated for the prevention embolic events (TIA's or CVA's).

Current articles are observational, and describe retrospectively the morbidity and mortality from atherosclerosis with aortic calcification.

the investigators assumption is that if aortic calcification is a marker for diffuse atherosclerosis, it has good correlation to criptogenous carotid artery disease, and can lead to early carotid artery disease evaluation and treatment.

Purpose - to find a reliable correlation between aortic calcification, and carotid artery stenosis (from atherosclerosis)

Method - two groups will be evaluated:

Group A - patients (age >40 years), that had a CT scan (chest/abdomen) for any indication, will be evaluated for aortic calcifications. The patients will be additionally examined for carotid artery stenosis by Doppler ultrasound. (100 patients) Group B - Patients that were diagnosed by Doppler ultrasound, and were found to have a severe carotid artery stenosis. These patients are scheduled for a computed tomography-angiography (regardless for the research) of the cervical arteries, will be additionally complete abdominal/chest tomography scan, without additional contrast. (50 patients).

Results - will be statistically evaluated - Group A - number of patients with aortic calcification, number of patients with carotid artery stenosis; Group B - Number of patients that have associated aortic calcification.

ELIGIBILITY:
Inclusion Criteria:

Group A - patients, age 40-99 years, that had a CT scan for any indication Group B - patients with severe carotid artery stenosis, that indicated for treatment

Exclusion Criteria:

* Group A - age <40 years
* Group B - carotid artery stenosis, without intention-to-treat

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group A - patients who had a CT scan Group B - patients who have severe carotid artery stenosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-02 (Estimated); Study Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Salamon, MD, Principal Investigator — Zim medical center; Alexander Altsuler, MD, Study Director — Ziv Medical Center